CLINICAL TRIAL: NCT03908502
Title: An Observational Study in Clinical Manifestations, Therapeutic Effects, Progress, and Prognosis of Radiotherapy-related Nervous System Complications
Brief Title: A Study in Radiotherapy-related Nervous System Complications
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yamei Tang, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: 20170601001
Record Dates: First submitted 2019-04-02; First posted 2019-04-09 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Nervous System Complication
Keywords: Radiotherapy; Nervous System Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Years
Biospecimen Retention: Samples With DNA — Blood sample are obtained in order to investigate significant genes, proteins and metabolites involved in the development and progress of radiotherapy-related nervous system complications. Genomics, metabolomics and proteomics are performed to detect potential genes, proteins and metabolites. Stool sample are obtained in order to investigate interactions between the gut microbiota, immune and nervous systems in radiotherapy-related nervous system complications. Cerebrospinal fluid (CSF) or biopsy samples are obtained if needed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose: This observational study aims to evaluate the clinical manifestations, therapeutic effects, progress and prognosis in radiotherapy-related nervous system complications.

OUTLINE: This is an observational clinical trial. Patients are enrolled and administrated with optimized clinical treatment. Blood, urine, stool, cerebrospinal fluid (CSF), imaging and other examinations, and scale assessments are regularly performed to evaluate the state of the disease.

Further study details are provided by Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University/Yamei Tang.

Primary outcome measure: The primary endpoint is overall survival.

DETAILED DESCRIPTION:
BACKGROUND

Radiotherapy is a key component in the management of head and neck tumors and primary or metastatic cancer of the central nervous system. Various radiation treatment methods employ different types of fractionation and conformational protocols designed to deliver focused radiation to target regions to maximize the lethal effect on the neoplasm and minimize the extraneous dose on normal brain tissue and other adjacent organs at risk. The outcomes of these clinical protocols may be complicated by radiation effects on normal brain parenchyma and other nervous system, resulting in a spectrum of phenotypes that range from clinically asymptomatic changes to radiotherapy-related nervous system complications with severe neurological defects, including delayed radiation-induced brain necrosis, myelopathy and nerve injury.

STUDY DESIGN:

Interventions Patients are enrolled and administrated with optimized clinical treatment.

Follow-up examinations

1. Blood, urine and stool examinations, such as biochemical A, coagulation routine, thyroid function, EB virus DNA, erythrocyte sedimentation rate, morning cortisol, urine sodium and potassium, gonadal hormone, growth hormone, glycosylated hemoglobin.
2. Imaging examinations, such as MR, CT, ultrasound. X ray is performed if needed.
3. Other examinations, such as pure tone audiometry, fundus exam, visual exam, VEP, OCTA, visual field exam.
4. Scale assessments about neurological function, radiation injury, common psychiatric disorders, cognitive function, quality of life, drug side effect, sleep and pain, such as LENT/SOMA, WHO-QOL, MoCA, MMSE, Hamilton anxiety scale, Hamilton depression scale, Pain numerical rating scale, Drug side effect scale, ADAS-cog, fatigue self-assessment scale (FSAS), Neuropsychiatric Inventry (NPI) total score, Clinical Dementia Rating Scale, Barthel index, UPDRS, Self-Rating Scale of Sleep (SRSS), NCI-CTCAE, CIBIC-plus and SSA.
5. Blood sample are obtained in order to investigate significant genes, proteins and metabolites involved in the development and progress of radiotherapy-related nervous system complications. Genomics, metabolomics and proteomics are performed to detect potential genes, proteins and metabolites. Stool sample are obtained in order to investigate interactions between the gut microbiota, immune and nervous systems in radiotherapy-related nervous system complications. Cerebrospinal fluid (CSF) and biopsy samples are obtained if needed.

ELIGIBILITY:
Inclusion Criteria

* Receipt of radiotherapy

Exclusion Criteria

* Inability to sign a written informed consent.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Radiotherapy is a key component in the management of head and neck tumors and primary or metastatic cancer of the central nervous system. The outcomes of various radiation protocols may be complicated by radiation effects on normal brain parenchyma and other nervous system, resulting in a spectrum of phenotypes that range from clinically asymptomatic changes to radiotherapy-related nervous system complications with severe neurological defects, including delayed radiation-induced brain necrosis, myelopathy and nerve injury.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2037-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Baseline until death or up to Year 20
  Overall survival is the duration between the first day of study enrollment to death. For participants who are alive, overall survival is censored at the last contact.

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, M.D., PhD., Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li H, Rong X, Hu W, Yang Y, Lei M, Wen W, Yue Z, Huang X, Chua MLK, Li Y, Cai J, He L, Pan D, Cheng J, Pi Y, Xue R, Xu Y, Tang Y. Bevacizumab Combined with Corticosteroids Does Not Improve the Clinical Outcome of Nasopharyngeal Carcinoma Patients With Radiation-Induced Brain Necrosis. Front Oncol. 2021 Sep 28;11:746941. doi: 10.3389/fonc.2021.746941. eCollection 2021. PMID 34650930